CLINICAL TRIAL: NCT03078894
Title: A Pilot Study Examining for the Presence of Fecal Coliforms in Peruvian Water Sources and the Association of Tropical Diseases Within Peru
Brief Title: A Pilot Study Examining for the Presence of Fecal Coliforms and Tropical Diseases in Peru
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: BioRed LLC (Other)
Responsible Party: Sponsor
Other Study IDs: CUIRBTL231
Record Dates: First submitted 2017-03-08; First posted 2017-03-14 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Tropical Disease
Keywords: Zika; Dengue; Chikagunya; Peru
MeSH Terms: conditions — Zika Virus Infection; Dengue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Districts: Contaminated Water: Subjects in this group are from districts that have contaminated water sources.
  Interventions: Diagnostic Test: Zika; Diagnostic Test: Chikagunya; Diagnostic Test: Dengue
- Districts: Uncontaminated Water: Subjects in this group are from districts that do not have contaminated water sources.
  Interventions: Diagnostic Test: Zika; Diagnostic Test: Chikagunya; Diagnostic Test: Dengue

INTERVENTIONS:
Diagnostic Test: Zika — Zika Diagnostic test
Diagnostic Test: Chikagunya — Chikagunya Diagnostic test
Diagnostic Test: Dengue — Dengue Diagnostic test

SUMMARY:
Tropical diseases are continuously on the rise throughout the world as they are spreading and manifesting in various locations globally. The more prominent vector tends to be the mosquito after it bites a previously infected host. The viruses of Zika, Chikungunya, and Dengue are some of the tropical diseases that are affecting large populations and expanding rapidly. Developing countries are at the highest risk because of the lack of preventive methods that are customarily demonstrated in developed countries. Sanitation issues complicate the problem as contaminated wastewater is ideal for mosquitos to lay eggs. In addition, the organic material in the wastewater serve as food for larvae. The purpose of this study is to test bodies of waters in Peru and examine if contaminated water is a contributing factor in the proportion of the population infected with Zika, Chikanguyna or Dengue.

DETAILED DESCRIPTION:
Tropical diseases are active in South America and measures need to be taken to control these diseases. Sanitation is a major contributing factor as it serves for an ideal breeding ground for vectors. The EPA regulates water contamination and states that a water source can be recognized as contaminated if it contains anything above zero total coliforms. The severity of the water contamination within Peru can be observed by the presence of thermotolerant coliforms in 48% of all water samples. Studies have also found that on 23% of hands, 16% of utensils, and 4% of meals, E. coli was present. The most frequently contaminated item was kitchen cloths in which 89% had coliforms and 42% with E. coli. In 33% of drinking water, 27% of meals, and 23% kitchen utensils, diarrheagenic E. coli was present.

The purpose behind the research being conducted is to assist Peru concerning various factors in order to facilitate the process of working towards the reduction or complete elimination of tropical disease infections such as Dengue, Zika, and Chikungunya. The reason Peru has been identified as being the focal point for the proposed research lies within the factors that surround Peru. Peru is considered a developing country and with that encompasses consequential issues. These issues can manifest in malnutrition, disease ridden environments, debilitating physical repercussions, and many other linked issues.5 Peru also has a substantial market in which producers partake in sugar cane cultivation. "In Peru, Maple Energy anticipates that in 2013, it will harvest 1.075 million gross tons of sugar cane from its plantation for ethanol production." This is significant considering that sugar cane and molasses production attracts mosquitoes and creates a prime nesting ground for mosquitos considering the product as well as the climate which is required to grow these items. The fact that Dengue is so rampant in Peru presents the great possibility that the masking of other infections with similar symptoms such as Chikungunya and Zika is present. Given that Peru is a developing country makes this fact even more feasible considering the minimal access to quality healthcare in many locations, especially rural communities. The location of Peru gives rise to believe that many patients go undiagnosed or misdiagnosed since Peru borders Brazil, in which currently Zika and Chikungunya are currently epidemics sweeping the country. The lack of mandated hygienic practices allows the circulation of many diseases to fester and plague the Peruvian society.

ELIGIBILITY:
Inclusion Criteria:

* From the Following Districts: Tuman, Pomalca, Patapo, Pimentel
* Over the age of 18

Exclusion Criteria:

* Not currently taking antiviral or antimicrobial medication

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Residents living in Tuman, Pomalca, Patapo and Pimentel that are over the age of 18 will be selected at random to participate in this study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-03-17 (Actual); Primary Completion 2017-05-01 (Estimated); Study Completion 2017-05-01 (Estimated)

PRIMARY OUTCOMES:
The number of contaminated water bodies | March 20th - April1st
  This is the number of contaminated water sources with fecal coliform

SECONDARY OUTCOMES:
Proportion of population with Zika, Dengue or Chikagunya infections | March 20th - May 1st
  The proportion of people that are positive for Zika, Dengue or Chikagunya infections

CONTACTS AND LOCATIONS:
Overall Officials: Trentice Lazard, Principal Investigator — Campbell University
Locations (4):
- Peru (4):
  - BioRed, Hacienda Pucala, Lambayeque
  - BioRed, Pátapo, Lambayeque
  - BioRed, Tumán, Lambayeque
  - BioRed, Pomalca

IPD SHARING:
Plan to Share IPD: Undecided